CLINICAL TRIAL: NCT02010333
Title: A Pediatric Safety and Pharmacokinetic Study of Ha44 Gel Administered Topically for the Treatment of Head Lice Infestation
Brief Title: A Pediatric Safety and Pharmacokinetics Study of Ha44 Gel Administered Topically for Treatment of Head Lice Infestation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ha03-003
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Head Lice Infestation
MeSH Terms: interventions — Benzyl Alcohol

ARMS (1):
- Ha44 Gel 0.74% w/w (Experimental): Open label, one arm
  Interventions: Drug: Ha44 Gel 0.74% w/w

INTERVENTIONS:
Drug: Ha44 Gel 0.74% w/w — HA44 Gel 0.74% comprises of Abametapir as the active pharmaceutical ingredient and Benzyl Alcohol as one of the excipients.
  Other Names: Abametapir 0.74%; Benzyl Alcohol

SUMMARY:
The primary purpose of the study is to evaluate safety and tolerability of a single application of Ha44 Gel 0.74% w/w for the treatment of head lice. Secondary purpose is to evaluate PK of Ha44 and benzyl alcohol under conditions of maximal exposure in pediatric population.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 6months < 3years of age
2. Good health
3. Active head lice infestation defined as the presence of at least 3 live lice
4. Dermatological condition of scalp (at least G2 erythema or pruritus with evidence of excoriation/inflammation)
5. Parent/guardian agrees to allow PK samples collected
6. Signed Informed Consent Form

Exclusion Criteria:

1. Condition or illness that in the opinion of the investigator may interfere with the study results.
2. Current dermatological disease that may compromise the health of subject or the assessment of safety. Subjects with scalp ulceration or evidence of scalp infection should not be enrolled.
3. Prior reaction to product containing piperonyl butoxide, pyrethrin, or pyrethrum extract.
4. Receiving systemic or topical medication that may interfere the study results.
5. Received an investigational agent within 30 days prior to Day 0.

Ages: 6 Months to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2013-04; Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of Ha44 Gel | 8 months
  Clinically significant changes in Physical Examinations, vital signs, safety laboratory tests and assessments of scalp and eye irritation and Electrocardiogram. The frequency and severity of Adverse Events.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Universal Biopharma Research Institute, Dinuba, California
  - Axis Clinical Trials, Los Angeles, California